CLINICAL TRIAL: NCT04959981
Title: A Phase 1b Master Protocol of Agents Targeting the Mitogen-Activated Protein Kinase Pathway in Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: A Study of Anti-Cancer Therapies Targeting the MAPK Pathway in Patients With Advanced NSCLC
Acronym: HERKULES-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Erasca, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ERAS-007-02
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Advanced Non-squamous Non-small-cell Lung Cancer
Keywords: EGFR; epidermal growth factor receptor; mutation; biomarker; NSCLC; Tagrisso; osimertinib; ERK; MAPK; sotorasib; Lumakras; KRAS; G12C; SHP2; PTPN11; molecular alterations; Kirsten rat sarcoma; Non-small cell lung cancer; Lung neoplasms; Thoracic neoplasms; ERAS-601; ERAS-007
MeSH Terms: conditions — Noonan Syndrome; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Thoracic Neoplasms | interventions — osimertinib; sotorasib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation (Part 1): ERAS-007 plus osimertinib (Experimental): ERAS-007 will be orally administered in combination with osimertinib to study participants with EGFRm NSCLC in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007; Drug: Osimertinib
- Dose Escalation (Part 2): ERAS-007 plus sotorasib (Experimental): ERAS-007 will be orally administered in combination with sotorasib to study participants with KRAS G12Cm NSCLC in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-007; Drug: Sotorasib
- Dose Escalation (Part 3): ERAS-601 plus sotorasib (Experimental): ERAS-601 will be orally administered in combination with sotorasib to study participants with KRAS G12Cm NSCLC in sequential ascending doses until unacceptable toxicity, disease progression, or withdrawal of consent.
  Interventions: Drug: ERAS-601; Drug: Sotorasib
- Dose Expansion (Part 4): ERAS-007 plus osimertinib (Experimental): ERAS-007 will be orally administered at the recommended dose (as determined from Part 1) in combination with osimertinib to study participants with EGFRm NSCLC.
  Interventions: Drug: ERAS-007; Drug: Osimertinib
- Dose Expansion (Part 5): ERAS-007 plus sotorasib (Experimental): ERAS-007 will be orally administered at the recommended dose (as determined from Part 2) in combination with sotorasib to study participants with KRAS G12Cm NSCLC.
  Interventions: Drug: ERAS-007; Drug: Sotorasib
- Dose Expansion (Part 6): ERAS-601 plus sotorasib (Experimental): ERAS-601 will be orally administered at the recommended dose (as determined from Part 3) in combination with sotorasib to study participants with KRAS G12Cm NSCLC.
  Interventions: Drug: ERAS-601; Drug: Sotorasib

INTERVENTIONS:
Drug: ERAS-007 — Administered orally
  Arms: Dose Escalation (Part 1): ERAS-007 plus osimertinib; Dose Escalation (Part 2): ERAS-007 plus sotorasib; Dose Expansion (Part 4): ERAS-007 plus osimertinib; Dose Expansion (Part 5): ERAS-007 plus sotorasib
Drug: ERAS-601 — Administered orally
  Arms: Dose Escalation (Part 3): ERAS-601 plus sotorasib; Dose Expansion (Part 6): ERAS-601 plus sotorasib
Drug: Osimertinib — Administered orally
  Other Names: Tagrisso
  Arms: Dose Escalation (Part 1): ERAS-007 plus osimertinib; Dose Expansion (Part 4): ERAS-007 plus osimertinib
Drug: Sotorasib — Administered orally
  Other Names: Lumakras
  Arms: Dose Escalation (Part 2): ERAS-007 plus sotorasib; Dose Escalation (Part 3): ERAS-601 plus sotorasib; Dose Expansion (Part 5): ERAS-007 plus sotorasib; Dose Expansion (Part 6): ERAS-601 plus sotorasib

SUMMARY:
* To evaluate the safety and tolerability of escalating doses of ERAS-007 or ERAS-601 in combination with other cancer therapies in study participants with advanced non-small cell lung cancer (NSCLC).
* To determine the Maximum Tolerated Dose (MTD) and/or Recommended Dose (RD) of ERAS-007 or ERAS-601 administered in combination with other cancer therapies.
* To evaluate the antitumor activity of ERAS-007 or ERAS-601 in combination with other cancer therapies.
* To evaluate the PK profiles of ERAS-007 or ERAS-601 and other cancer therapies when administered in combination.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, multicenter master protocol evaluating safety, tolerability, and antitumor activity of ERAS-007 or ERAS-601 in combination with other cancer therapies in study participants with advanced NSCLC. The study will commence with the following dose escalation cohorts: ERAS-007 plus osimertinib in study participants with advanced NSCLC harboring epidermal growth factor receptor-sensitizing mutation(s) (EGFRm); ERAS-007 or ERAS-601 plus sotorasib in study participants with advanced NSCLC harboring Kirsten rat sarcoma G12C mutation (KRAS G12Cm). Dose expansion will follow and will evaluate ERAS-007 or ERAS-601 drug combinations administered at the RD identified from each respective dose escalation cohort in study participants with advanced EGFRm or KRAS G12Cm NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Willing and able to give written informed consent.
* Have histologically or cytologically confirmed NSCLC, with presence of EGFR mutation(s) sensitive to EGFR inhibitors, or KRAS G12C mutation.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Adequate bone marrow and organ function.
* Have ECOG performance status of 0 or 1.
* Willing to comply with all protocol-required visits, assessments, and procedures.
* Able to swallow oral medication.

Exclusion Criteria:

* Concurrent treatment with any systemic anticancer therapy for NSCLC, including any approved or investigational agent.
* For participants with EGFRm NSCLC: prior therapy with a RAS, RAF, MEK, or ERK inhibitor.
* For participants with KRAS G12Cm NSCLC: prior therapy with a SHP2, ERK, or KRAS G12C inhibitor (depending on which cohort is being considered for enrollment).
* Palliative radiotherapy within 7 days of enrollment.
* History of unacceptable toxicity to treatment with osimertinib or sotorasib.
* Major surgery within the 28 days of enrollment.
* Unresolved toxicities from prior systemic therapy greater than NCI CTCAE grade 1 at time of enrollment, except for toxicities not considered a safety risk (eg, alopecia, vitiligo, and grade 2 neuropathy due to prior chemotherapy).
* History of another malignancy ≤5 years prior to first dose, except for patients who are disease-free for >2 years after treatment with curative intent or who have carcinoma in situ.
* Symptomatic and unstable brain metastases, or spinal cord compression, except for patients who have completed definitive therapy (surgery or radiotherapy), are not on steroids, and have a stable neurologic status for a least 2 weeks after completion of the definitive therapy and steroids.
* History of or clinically active ILD, drug induced ILD, or radiation pneumonitis that required steroid treatment.
* Impaired cardiovascular function or clinically significant cardiovascular disease.
* History or current evidence of retinal pigment epithelial detachment (RPED), central serous retinopathy, retinal vein occlusion (RVO), or predisposing factors to RPED or RVO.
* Any evidence of severe or uncontrolled systemic disease or evidence of any other significant clinical disorder or laboratory finding that renders the patient inappropriate to participate in the study.
* Pregnant or breastfeeding women.
* Contraindication to osimertinib or sotorasib use as per local label.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) | Study Day 1 up to Day 22
  Based on adverse events observed
Maximum Tolerated Dose (MTD) | Study Day 1 up to Day 22
  Based on adverse events observed
Recommended Dose (RD) | Study Day 1 up to Day 22
  Based on adverse events observed
Adverse Events | Assessed up to 24 months from time of first dose
  Incidence and severity of treatment-emergent AEs and serious AEs

SECONDARY OUTCOMES:
Plasma concentration (Cmax) | Study Day 1 up to Day 22
  Maximum plasma concentration of ERAS-007 or ERAS-601 and other cancer therapies
Time to achieve Cmax (Tmax) | Study Day 1 up to Day 22
  Time to achieve maximum plasma concentration of ERAS-007 or ERAS-601 and other cancer therapies
Area under the curve | Study Day 1 up to Day 22
  Area under the plasma concentration-time curve of ERAS-007 or ERAS-601 and other cancer therapies
Half-life | Study Day 1 up to Day 22
  Half-life of ERAS-007 or ERAS-601 and other cancer therapies
Objective Response Rate (ORR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1
Duration of Response (DOR) | Assessed up to 24 months from time of first dose
  Based on assessment of radiographic imaging per RECIST version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Antal, Study Director — Senior Director, Clinical Development
Locations (11):
- United States (11):
  - City of Hope, Duarte, California
  - UC Irvine, Chao Family Comprehensive Cancer Center, Orange, California
  - UC Los Angeles, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Research Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Hackensack University Medical Center (John Theurer Cancer Center), Hackensack, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute (Tennessee Oncology), Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No